CLINICAL TRIAL: NCT02191475
Title: Tigecycline (Hai Zheng Li Xing®) Combined With Piperacillin/Tazobactam (Tazocin ®) Empirical Treatment of Severe Sepsis and Septic Shock in Patients With Abdominal Infection
Brief Title: Effect Study of Tigecycline to Treat Severe Sepsis and Septic Shock
Acronym: Tigecycline
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WDH2014
Record Dates: First submitted 2014-06-24; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-05

CONDITIONS: Abdominal Infection
Keywords: sepsis shock; Tigecycline; Piperacillin / tazobactam; Abdominal infection
MeSH Terms: conditions — Intraabdominal Infections | interventions — Glycopeptides; Carbapenems; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glycopeptide plus carbapenem (Active Comparator): The control group antibiotic selection according to the classical scheme use of glycopeptide plus carbapenem antibiotic (or oxazolidinone antibiotics), with or without antifungal therapy, dose of imipenem/cilastatin 500mg, IVdrip, 3~4 times/d, or meropenem 1g, IVdrip, 3 times/d; vancomycin for 15mg/kg,2 times/d, or linezolid 300mg, IVdrip, 2 times/d; these drugs are required to state organ function in patients with drug doses adjustment, treatment for 3-5 days.
  Interventions: Drug: glycopeptide plus carbapenem
- Haizheng Li Xing ® plus tazocin ® (Experimental): Tigecycline (Haizheng Li Xing ®) combined with piperacillin / tazobactam (tazocin ®), with or without antifungal therapy, dose of tigecycline first dose 100 mg, 50 mg, every 12 hours, piperacillin / tazobactam 4.5g, ivdrip, 3-4 times a day, each time the infusion of 3 hours, treatment for 3-5 days.
  Interventions: Drug: Haizheng Li Xing ® plus tazocin ®

INTERVENTIONS:
Drug: glycopeptide plus carbapenem — The control group antibiotic selection according to the classical scheme use of glycopeptide plus carbapenem antibiotic (or oxazolidinone antibiotics), with or without antifungal therapy
  Other Names: The clinical curative effect
  Arms: glycopeptide plus carbapenem
Drug: Haizheng Li Xing ® plus tazocin ® — Tigecycline (Haizheng Li Xing ®) combined with piperacillin/tazobactam (tazocin ®), with or without antifungal therapy
  Other Names: The clinical curative effect
  Arms: Haizheng Li Xing ® plus tazocin ®

SUMMARY:
Selection of tigecycline in severe sepsis and septic shock patients in empirical antibiotic therapy (Hai Zheng Energy Star ®) combined with piperacillin / tazobactam (tazocin ®) scheme, compared with the classical scheme, evaluate its efficacy, safety index.

DETAILED DESCRIPTION:
Tigecycline as representative glycylcycline antibiotics, has wide antibacterial spectrum and strong antibacterial activity, tigecycline in almost all of the gram positive bacteria and most gram negative bacteria and atypical pathogens, anaerobic bacteria are very good antibacterial activity except Pseudomonas aeruginosa, Proteus. Safety on organ function, in patients with renal insufficiency or in dialysis patients, no dose adjustment is required application of tigecycline, mild to moderate hepatic insufficiency patients do not need to adjust the dose of tigecycline. Piperacillin / tazobactam also is a broad spectrum, potent antibiotics, especially strong bactericidal activity against Pseudomonas aeruginosa, including resistant enzyme producing gram negative bacilli, in accordance with its pharmacokinetic pharmacodynamic characteristics of prolonged infusion time can obtain a stronger bactericidal activity. These two potent drugs have broad antimicrobial spectrum, strong bactericidal activity, and provide for the treatment of severe sepsis and septic shock a new choice in antibiotic selection, to a certain extent reduces the resistance pressure, and have more clinical safety.

ELIGIBILITY:
Inclusion Criteria:

* Be consistent with severe sepsis and septic shock diagnosis standards
* Age above 18 years old, is expected in more than 5 days in ICU
* APACHEⅡ score>15
* By the patients themselves or their authorized person agreed to participate in the clinical trial and signed the informed consent

Exclusion Criteria:

* Allergic to penicillin, or of tigecycline allergic patients
* Patients with abnormal liver function is severe
* Be pregnant or lactating women
* Be not signed the informed consent of patients
* Any can be expected to increase patient risk or other factors can interfere with the results of a clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment between Tigecycline plus tazocin and classic anti infection method | 2 weeks
  Two groups of patients were assessed anti infection treatment effect per day. Including: temperature, procalcitonin, blood routine, liver and kidney function, bacteriological evidence, hemodynamics
  Effects of Haizheng Li Xing ® combined with tazocin ® in clinical treatment is not inferior to the classical antibiotics scheme

SECONDARY OUTCOMES:
Successful rate between two groups with abnormal renal function and liver function abnormalities which should adjust dose of drugs | 2 weeks
  Evaluation of two groups of patients EGDT treatment compliance rate, mortality rate (the success rate of treatment), ICU stay time.

OTHER OUTCOMES:
Residence time and expenses in ICU | 2 weeks
  Patients with ICU residence time and expenses have no difference between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Donghao, Chief, Study Chair — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- TianjinCIH, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Background] Sartelli M, Catena F, Coccolini F, Pinna AD. Antimicrobial management of intra-abdominal infections: literature's guidelines. World J Gastroenterol. 2012 Mar 7;18(9):865-71. doi: 10.3748/wjg.v18.i9.865. PMID 22408344
- [Result] Eckmann C, Montravers P, Bassetti M, Bodmann KF, Heizmann WR, Sanchez Garcia M, Guirao X, Capparella MR, Simoneau D, Dupont H. Efficacy of tigecycline for the treatment of complicated intra-abdominal infections in real-life clinical practice from five European observational studies. J Antimicrob Chemother. 2013 Jul;68 Suppl 2:ii25-35. doi: 10.1093/jac/dkt142. PMID 23772043
- [Result] Hawkey P, Finch R. Tigecycline: in-vitro performance as a predictor of clinical efficacy. Clin Microbiol Infect. 2007 Apr;13(4):354-62. doi: 10.1111/j.1469-0691.2006.01621.x. PMID 17359318